CLINICAL TRIAL: NCT04406987
Title: Degenerative Segmental Instability in Lumbar Spinal Stenosis Patients - Study on Instability, Clinical Outcomes, Reoperation Rate With a 2 Year Follow up
Brief Title: Instability in the Lumbar Spine of Patients With Age Related Changes and Narrowing of the Spinal Canal (Spinal Stenosis)
Status: Completed | Type: Observational
Sponsor: Spine Centre of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: 20/7176; 20202000-22 (Other: National Committee on Health Research Ethics)
Record Dates: First submitted 2020-05-24; First posted 2020-05-29 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Degenerative Spondylolisthesis
Keywords: instability; anterior translation; slip; segmental motion; radiologic assesment; lumbar MRI; MRI characteristics
MeSH Terms: interventions — Decompression; Gene Fusion; Arthrodesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- decompression: patients treated with decompression for lumbar spinal stenosis
  Interventions: Procedure: decompression
- fusion: patients treated with decompression with fusion for lumbar spinal stenosis
  Interventions: Procedure: fusion

INTERVENTIONS:
Procedure: decompression — surgical technique for neural decompression varied based on surgeon's preference, but always with preservation for spinous processes. Either open with or without microscope or using tubular retractors.
  Groups: decompression
Procedure: fusion — fusion techniques consisted besides decompression of additional implantation of pedicle screws with rods, with or without intervertebral fusion and cage(s). Non-instrumented technique with allograft bone. Fusion technique on surgeon's discretion.
  Other Names: arthrodese
  Groups: fusion

SUMMARY:
Age related changes in the lumbar spine can lead to narrowing of the spinal canal (spinal stenosis) causing leg and back pain. Spinal stenosis can be associated with a misalignment of the spine caused by forward slippage of a vertebrae over another. This instability is diagnosed using diagnostic imaging. With signs of instability the spine surgeon might choose a fusion of the vertebrae. This is a more complex procedure in relation to the simple decompression preformed without instability for spinal stenosis.

The purpose of this study is to identify characteristics of instability of the lumbar spine on diagnostic imaging, and investigate associations with surgical data and patient reported outcomes from the National Spine databases from Denmark and Sweden.

This will support spine surgeons in providing evidence-based surgical treatment for spinal stenosis with or without signs of instability

DETAILED DESCRIPTION:
A multicenter retrospective cohort study of prospectively collected data from national spine surgery databases in Denmark and Sweden. This project is a collaboration between sector for spine surgery and research Middelfart Hospital and spine surgeons at Orebro Hospital and Lund Hospital in Sweden.

Data subtracted from Danish national spine surgery database, DaneSpine, from Middelfart Hospital, and Swedish Spinal Register, SweSpine, from hospitals in Malmö, Lund, Trelleborg and Karlskroga.

Both databases are clinical quality databases with a high response-rate. DaneSpine is administered by Danish Society of Spine Surgeons and is managed by secretary of DaneSpine. SweSpine is administered by Swedish Society of Spinal Surgeons and managed

Patients are invited to register when scheduled for surgery. Patients signs informed consent and receives follow-up questionaires 3 and 6 months, one, two, 5 and 10 years post-surgery. Questionaires are validated PROM (patient reported outcome measures) and PREM (patient reported experience measures).

The surgeon is responsible for registering surgical data, including complications and reoperations.

Data relevant for present study will be applied for at the respective societies and managed and stored in compliance with General Data Protection Regulation.

The EasyWiz software (Medical Insight, Chicago, IL, USA) is used for analysis of all MRIs and radiographs.

All imaging will be analyzed by 2 independent examiners. The interobserver reliability will be calculated.

Missing data such as variables reported as missing or non-reported will not be included in statistical analysis.

Statistics: significance of difference in mean values between groups for continuous normally distributed data unpaired t-test. Categorical variables normally distributed: Chi-squared/Fishers exact test. Multivariable regression analysis. Kappa statistics for interobserver reliability presented in the article.

ELIGIBILITY:
Inclusion Criteria:

- MRI verified spinal stenosis patients with or with out degenerative spondylolisthesis (> 3mm anterior translation in lumbar MRI), who underwent surgery at L4/L5 level with either decompression alone or decompression with fusion between 2010 and 2017. Included ICD-10 diagnostic groups DM480 and DM431. Must have standing lateral radiographs preoperatively. Completed 2 year follow up.

Exclusion Criteria:

* previous surgery at the same level,
* malignancy or undergoing treatment for malignancy
* scoliosis Cobb angel >20 degrees

Ages: 18 Years to 110 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with symptomatic, MRI-verifeis lumbar spinal stenosis referred to Spine Center of Southern Denmark between 2010-2017. And same study population referred to Spine Centers at hospitals in Malmö, Lund, Trelleborg and Karlskroga Sweden between 2010-2017.
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
facet joint gap | pre-surgery
  MRI proxies 1

SECONDARY OUTCOMES:
facet angel | pre-surgery
  MRI proxies 2
disc height | pre-surgery
  MRI proxies 3
anterior translation | pre-surgery
  MRI proxies 4
intradiscal vacuum | pre-surgery
  MRI proxies 5
radiographic slip | pre-surgery
  anterior translation on lateral radiograph

OTHER OUTCOMES:
VAS leg | pre-surgery and 3 months, 12 months and 2 years post-surgery
  Visual Analog Scale (VAS) a 0 (no pain) to 100 (severe pain) point scale
VAS back | pre-surgery and 3 months, 12 months and 2 years post-surgery
  Visual Analog Scale (VAS) a 0 (no pain) to 100 (severe pain) point scale
EQ-5D | pre-surgery and 3 months, 12 months and 2 years post-surgery
  EuroQol (EQ-5D) measures health-related quality of life on a scale where 0.0 equal's death and 1.0 equals perfect health
ODI | pre-surgery and 3 months, 12 months and 2 years post-surgery
  Oswestry Disability Index (ODI) questionnaire scores range from 0 (no disability) to 100 (total disability)
patient characteristics | pre-surgery and 3 months, 12 months and 2 years post-surgery
  age, gender, BMI, smoking, diabetes
reoperation | 3 months, 12 months and 2 years post-surgery
  operation on index level after primary operation and discharge within follow-up period
complication | during surgery or during admission
  perisurgical complication within admission.

CONTACTS AND LOCATIONS:
Overall Officials: Signe Forbech Elmose, M.D., Principal Investigator — Spine Center of Southern Denmark, Lillebaelt Hospital, Denmark
Locations (1):
- Center for spine surgery and research, Spine Center of Southern Denmark, Middelfart, Denmark

IPD SHARING:
Plan to Share IPD: No